CLINICAL TRIAL: NCT07363161
Title: BASel Kosten-Effektivitäts-Trial: Drug-coated BALLoon vs. Drug-eluting Stent Strategy in High-risk Patients With Coronary Artery Disease
Brief Title: Drug-coated Balloon (DCB) vs. Drug-eluting Stent (DES) in High-risk Patients With Coronary Artery Disease (CAD)
Acronym: BASKET BALL
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: B. Braun Melsungen AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AAG-G-H-24094
Record Dates: First submitted 2026-01-15; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Coronary Artery Disease (CAD)
Keywords: CAD; SCB; SeQuent® SCB
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SeQuent® SCB-based strategy (Active Comparator): all target lesions should be treated with the SeQuent® SCB after adequate lesion preparation. If the angiographic result is unacceptable following lesion preparation or after DCB treatment (e.g., flow-limiting dissection or residual stenosis >30%), additional therapeutic steps should be considered.
  For non-left main bifurcation lesions, if the side branch requires treatment, it should also be treated with the SeQuent® SCB after adequate lesion preparation. If an unacceptable angiographic result, defined as >70% residual stenosis or major recoil at the side branch ostium, is obtained, or if there is an imminent risk of vessel compromise, further therapeutic steps are required. Those steps may include optimized lesion preparation to avoid DES implantation; however, DES may be implanted if all other attempts fail.
  Interventions: Device: PCI
- DES-based strategy (Active Comparator): all target lesions should be treated with DES. The use of DCB in the DES arm is strongly discouraged. If DES delivery is not feasible due to anatomical or other reasons, the operator may consider alternative treatments, such as more deliverable DES or plain old balloon angioplasty (POBA), while keeping the patients in the DES group. In case of bifurcation treatment, both DES and POBA are allowed.
  Any use of DCB in the DES arm shall be justified.
  Interventions: Device: PCI

INTERVENTIONS:
Device: PCI — PCI with SeQuent® SCB
  Arms: SeQuent® SCB-based strategy
Device: PCI — PCI with DES
  Arms: DES-based strategy

SUMMARY:
The main objective of this randomized, multicenter, international, open-label clinical trial is to demonstrate that, in the context of percutaneous coronary intervention for complex coronary artery disease, a SeQuent® SCB interventional strategy is non-inferior to a new-generation

DES strategy in terms of a 12- and 36-month composite of Target Vessel Failure (TVF), that includes:

* cardiovascular death (CV death),
* target vessel related MI (TV-MI),
* clinically indicated target vessel revascularization (ci-TVR),
* bleeding according to Bleeding Academic Research Consortium (BARC) Types 3-5.

Eligible subjects will be assigned in a 1:1 ratio to receive treatment of all lesions with either the SeQuent® SCB-based strategy or a DES-based strategy. The randomization will be performed prior to the index procedure once signed informed consent has been obtained and all eligibility criteria have been confirmed.

All Subjects will be followed for clinical outcomes at 3 months, 1, 2, and 3 years. A subset of 138 randomized patients will undergo control angiography after one-year clinical follow-up (+1 month). An independent core laboratory will analyze all baseline angiograms.

If, at 36 months, the non-inferiority of the SeQuent® SCB strategy compared to the DES strategy is achieved, superiority in terms of TVF and BARC Type 3-5 bleeding will be tested.

An optional extension of follow-up to 6 years may be implemented based on interim results and the joint decision of the Steering Committee and the Sponsor. Details regarding this optional extension are provided in the Clinical Investigation Plan.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be 18 years of age or older
* Subject can understand risks, benefits, and treatment alternatives of receiving DCB treatment or DES and provide written informed consent before any study-related procedure
* Subject should have a documented angina pectoris or silent ischemia as assessed by non-invasive testing, or functional invasive assessment, or equivalent (dyspnea, arrhythmia, ≥75% diameter stenosis without stress test at staged procedure), or unstable angina, hemodynamically stable NSTEMI and STEMI more than 48 hours after primary PCI and without residual thrombotic material
* Subject must be affiliated with a social security system, where applicable

Subject must have at least one of the high clinical or anatomical risk features:

High clinical risk, defined as:

* DM on treatment (insulin or oral antidiabetic agents), or
* At least 75 years of age, or
* CKD (eGFR <60 mL/min/1.73 m2), or
* Treated for ACS (unstable angina, hemodynamically stable NSTEMI, hemodynamically stable STEMI more than 48 hours after uneventful primary PCI and without residual thrombotic material), or
* High bleeding risk (defined by Academic Research Consortium criteria - ARC HBR)

OR

High anatomical risk lesions requiring treatment as follows:

* Multivessel treatment (two or three vessels)
* True bifurcation with side branch involvement
* Long lesions (≥36 mm)
* Lesion likely requiring calcium modification

In the case of multivessel (MV) disease, multiple vessels can be treated provided that all lesions are amenable to treatment with either DCB or DES and vessel size at the site of the lesion is >2.0 mm by visual assessment.

The trial does not restrict the number of target lesions. However, the operator should determine that all target lesions intended to be treated must be suitable for treatment with either DES or DCB. For patients randomized to the DCB arm, the likelihood of requiring provisional stenting must be assessed as less than 30% for each lesion requiring treatment.

Exclusion Criteria:

* Primary PCI (acute STEMI patients)
* Cardiogenic shock
* Subject enrolled in an active interventional trial
* Subject not able or unlikely to comply with the planned follow-ups
* Subject who is pregnant, nursing or planning to become pregnant during the study
* Subject not able to give informed consent
* Subject under judicial protection, guardianship or curatorship or patient deprived of their liberty by judicial or administrative decision (where applicable)
* Subject with a life expectancy <12 months
* Subjects with known allergies to antiplatelet agents (e.g., acetylsalicylic acid, P2Y12 inhibitors), anticoagulants (e.g., heparin, direct thrombin inhibitors), iodinated contrast media, or mTOR inhibitors (e.g., sirolimus and related compounds)
* Angiographic exclusion criteria:

  1. aorto-ostial lesions,
  2. coronary bypass grafts requiring intervention,
  3. chronic total occlusion requiring intervention
  4. Previous PCI at any time of a vessel intended to be treated (Instent-restenosis lesions excluded)
  5. Previous PCI within 30 days, except for recent STEMI, >48 hours after uneventful primary PCI and without residual thrombotic material on coronary angiography

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2184 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2031-03 (Estimated)

PRIMARY OUTCOMES:
Composite of Target Vessel Failure (TVF) and bleeding according to Bleeding Academic Research Consortium (BARC) Types 3-5 | at 12 months (after intervention)
Composite of TVF and bleeding BARC 3-5 | at 36 months

SECONDARY OUTCOMES:
Composite of TVF and bleeding BARC 3-5 | at 3 months
Composite of TVF and bleeding BARC 3-5 | at 24 months
Device-oriented Composite Endpoint (DOCE) | at 3 months
  a composite of cardiovascular death (CV death), device failure-related myocardial infarction (MI), and clinically indicated Target Lesion Revascularization (ci-TLR)
DOCE | at 12 months
DOCE | at 24 months
DOCE | at 36 months
TVF | at 3 months
TVF | at 12 months
TVF | at 24 months
TVF | at 36 months
Patient-oriented Composite endpoint (POCE) | at 3 months
  a composite of any death, any MI, any stroke, and any revascularization
POCE | at 12 months
POCE | at 24 months
POCE | at 36 months
Any death | at 3 months
Any death | at 12 months
Any death | at 24 months
Any death | at 36 months
CV death | at 3 months
CV death | at 12 months
CV death | at 24 months
CV death | at 36 months
Cardiac death | at 3 months
Cardiac death | at 12 months
Cardiac death | at 24 months
Cardiac death | at 36 months
Any MI | at 3 months
Any MI | at 12 months
Any MI | at 24 months
Any MI | at 36 months
Target Vessel-Related MI | at 3 months
Target Vessel-Related MI | at 12 months
Target Vessel-Related MI | at 24 months
Target Vessel-Related MI | at 36 months
Peri-procedural MI | at 3 months
  as defined by Drug Coated Balloon Academic Research Consortium (DCB ARC)
Peri-procedural MI | at 12 months
Peri-procedural MI | at 24 months
Peri-procedural MI | at 36 months
Spontaneous MI | at 3 months
  according to 4th Universal Definition of MI
Spontaneous MI | at 12 months
Spontaneous MI | 24 months
Spontaneous MI | at 36 months
BARC type ≥2 bleeding | at 3 months
BARC type ≥2 bleeding | at 12 months
BARC type ≥2 bleeding | at 24 months
BARC type ≥2 bleeding | at 36 months
BARC 3-5 bleeding | at 3 months
BARC 3-5 bleeding | at 12 months
BARC 3-5 bleeding | at 24 months
BARC 3-5 bleeding | at 36 months
Definite stent/lesion thrombosis | at 3 months
Definite stent/lesion thrombosis | at 12 months
Definite stent/lesion thrombosis | at 24 months
Definite stent/lesion thrombosis | at 36 months
Stroke | at 3 months
  ischemic and hemorrhagic
Stroke | at 12 months
Stroke | at 24 months
Stroke | at 36 months
Any TLR | at 3 months
Any TLR | at 12 months
Any TLR | at 24 months
Any TLR | at 36 months
ci-TLR | at 3 months
ci-TLR | at 12 months
ci-TLR | at 24 months
ci-TLR | at 36 months
Any TVR | at 3 months
Any TVR | at 12 months
Any TVR | at 24 months
Any TVR | at 36 months
ci-TVR | at 3 months
ci-TVR | at 12 months
ci-TVR | at 24 months
ci-TVR | at 36 months
Dual Antiplatelet Therapy (DAPT) burden | at 3 months
  total duration of DAPT and/or Single Antiplatelet Therapy (SAPT)
DAPT burden | at 12 months
DAPT burden | at 24 months
DAPT burden | at 36 months
Hospitalization related to study endpoints | at 3 months
Hospitalization related to study endpoints | at 12 months
Hospitalization related to study endpoints | at 24 months
Hospitalization related to study endpoints | at 36 months
Procedure success | at 3 months
  defined as Device success and freedom from in-hospital cardiovascular death, TLR, peri-procedural MI, any stroke, and BARC 3 or 5 bleeding
Procedure success | at 12 months
Procedure success | at 24 months
Procedure success | at 36 months
Device success (DCB) | at 3 months
  defined as successful delivery in time and inflation within 30-60 s of the allocated DCB device at the intended target lesion during an attempt with a DCB not previously used (first use); successful withdrawal of the device system; attainment of a final in-segment or in-lesion residual stenosis of <30% (except in the side branch ostium in nonleft main bifurcation lesions <70%) by visual estimate
Device success (DCB) | at 12 months
Device success (DCB) | at 24 months
Device success (DCB) | at 36 months
Device success (DES) | at 3 months
  defined as successful delivery, balloon expansion, and deployment of the first assigned DES at the intended target lesion; successful withdrawal of the device delivery system; attainment of a final in-stent residual stenosis of <20% by visual estimate
Device success (DES) | at 12 months
Device success (DES) | at 24 months
Device success (DES) | at 36 months
Metal burden | at 3 months
  by assessing the total stent length
Metal burden | at 12 months
Metal burden | at 24 months
Metal burden | at 36 months
In-segment net gain | assessed between 12 and 13 months
  Main angiographic endpoint after completion of the 12-month follow-up
Cost-effectiveness of DCB-based vs. DES-based strategy | at 12 months
Cost-effectiveness of DCB-based vs. DES-based strategy | at 24 months
Cost-effectiveness of DCB-based vs. DES-based strategy | at 36 months

CONTACTS AND LOCATIONS:
Locations (1):
- Stadtspital Zürich, Klinik für Kardiologie, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No